CLINICAL TRIAL: NCT01768247
Title: HCG Priming for Thin Endometrium in IVF
Brief Title: HCG (Human Chorionic Gonadotropin) Priming for Thin Endometrium in IVF (in Vitro Fertilization)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Human Reproduction & Genetics Foundation (Unknown)
Responsible Party: Principal Investigator, Papanikolaou Evangelos, MD,PHD, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THINENDOM001
Record Dates: First submitted 2013-01-12; First posted 2013-01-15 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Endometrial Thickness; Pregnancy Outcome
Keywords: endometrium; thickness; pregnancy; HCG; frozen cycles
MeSH Terms: interventions — Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HCG priming (Experimental): Patients in this arm after 7-9 days of estrogen replacement they will receive a 150 international units (IU) HCG every day for 7 days concomitantly with the estradiol
  Interventions: Drug: HCG (human chorionic gonadotropin)

INTERVENTIONS:
Drug: HCG (human chorionic gonadotropin) — 150 international units (IU) of HCG for seven days subcutaneously concomitantly with estrogens in preparation endometrium cycles fro frozen embryos replacement

SUMMARY:
A thin endometrium is one of the most difficult problems encountered in assisted reproduction every day practice Regarding the proliferative phase, several ways of treatment have been undertaken to circumvent thin endometrium trying to increase thickness with questionable results.

The objective of the current study will be whether a daily dose of 150 IU (international units) of human chorionic gonadotropin (HCG) for seven days concomitant with estrogen administration in estrogen replacement cycles can increase the endometrial thickness and improve pregnancy outcome.

DETAILED DESCRIPTION:
In this pilot study subjects with repeatedly resistant thin endometrium, less than 6mm, will be recruited. The investigators sought to investigate the possible role of adding low dose HCG in the follicular phase, on the endometrial growth and development. The investigators constructed this hypothesis based on the fact that LH/HCG (luteinizing hormone/human chorionic gonadotropin) receptor is present in endometrium and therefore a positive interaction could be anticipated when HCG is administered in the proliferative phase of endometrial growth. Furthermore, in a previous study, where human menopausal gonadotropin (hMG) -well known that renders its luteinizing hormone (LH) capacity due to low dose HCG contain- was compared to recombinant-follicular stimulating hormone (rec-FSH) during ovarian stimulation, endometrium was more likely to be iso-echogenic and hypo-echogenic in the hMG group, also anticipating a possible positive role of HCG activity.

ELIGIBILITY:
Inclusion Criteria:

* (1) Less than 6mm endometrial thickness before, (2) at least two failed implantations before

Exclusion Criteria:

* Abnormal uterine cavity in Hysteroscopy

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Endometrial thickness | 14 days after estrogen treatment
  measured by transvaginal ultrasound

SECONDARY OUTCOMES:
Pregnancy outcome | 5 weeks after embryotransfer
  Clinical pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Papanikolaou Evangelos, MD, Principal Investigator — HRG clinical director
Locations (1):
- HRG Foundation, Thessaloniki, Kalamaria, Greece

REFERENCES:
- [Background] Shufaro Y, Simon A, Laufer N, Fatum M. Thin unresponsive endometrium--a possible complication of surgical curettage compromising ART outcome. J Assist Reprod Genet. 2008 Aug;25(8):421-5. doi: 10.1007/s10815-008-9245-y. Epub 2008 Sep 17. PMID 18797990
- [Derived] Papanikolaou EG, Kyrou D, Zervakakou G, Paggou E, Humaidan P. "Follicular HCG endometrium priming for IVF patients experiencing resisting thin endometrium. A proof of concept study". J Assist Reprod Genet. 2013 Oct;30(10):1341-5. doi: 10.1007/s10815-013-0076-0. Epub 2013 Aug 16. PMID 23949214
- See also: Facility web page — http://www.hrg.gr